CLINICAL TRIAL: NCT04722224
Title: Home-based Pulmonary Rehabilitation in Patients With Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Polytechnic Institute of Porto (Other)
Collaborators: Nippon Gases Portugal (Unknown)
Responsible Party: Principal Investigator, Rui Vilarinho, Master, Polytechnic Institute of Porto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: reabilitar_DPOC_2
Record Dates: First submitted 2021-01-17; First posted 2021-01-25 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: COPD
Keywords: home-based pulmonary rehabilitation; exercise training; self-management
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention: Home-based pulmonary rehabilitation (Experimental): Patients will be treated for 12 weeks. The intervention consists in a strategic mixture of home visits and phone calls. The program includes exercise training and the self-management educational program Living Well with COPD.
  Interventions: Other: Home-based pulmonary rehabilitation

INTERVENTIONS:
Other: Home-based pulmonary rehabilitation — The reabilitAR program includes the self-management educational program Living Well with COPD. The exercise training will include endurance, resistance/strength, flexibility and balance training.

SUMMARY:
This project aims to assess the short-term effectiveness and responsiveness of a home-based pulmonary rehabilitation (PR) program (reabilitAR) in patients with chronic obstructive pulmonary disease (COPD). It is also an aim to establish the minimal clinically important differences for PR in patients with COPD for a novel incremental step test (exercise capacity outcome measure).

Patients will be recruited at hospitals. Sociodemographic, anthropometric, and comorbidities; vital signs and peripheral oxygen saturation; symptoms (dyspnea, fatigue); lung function; functional capacity; exercise capacity; the impact of the disease, balance, and cognitive function will be collected before the reabilitAR program. Additionally, health care utilization will be registered. Then, patients will be entered into the reabilitAR program (12 weeks). The intervention consists in a strategic mixture of home visits and phone calls. The program includes exercise training and the self-management educational program Living Well with COPD. After 12 weeks all outcome measures will be reassessed.

It is expected that the home-based approach will express benefits and reflect the concerns to provide appropriate responses to the patient's needs by increasing access to PR.

DETAILED DESCRIPTION:
The World Health Organization (WHO) indicates that hundreds of millions of people worldwide are affected by chronic respiratory diseases (CRD), including chronic obstructive pulmonary disease (COPD). Pulmonary rehabilitation (PR) is an essential component in the management of CRD with the aim to improve patients' exercise and functional capacity and psychological condition with long-term adherence to health-enhancing behaviors, including exercise training and self-management skills.

However, despite the well-known evidence, this service is mostly underutilized due to poor accessibility, with only 1% of worldwide availability of PR services for COPD patients. Thus, is important to undertake actions that improve access to and delivery of PR services for suitable patients. One of the strategies in the international guidelines is the creation of new models of programs, where a home-based approach is indicated.

The aim of this project is to assess the short-term effectiveness and responsiveness of a home-based pulmonary rehabilitation program (reabilitAR) in patients with COPD. It is also an aim to establish the minimal clinically important differences for PR in patients with COPD for a novel incremental step test (exercise capacity outcome measure).

The plan is to recruit the maximum of patients with COPD via clinicians at hospitals. This study will enroll adult patients with COPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria.

Patients will be referred by pulmonologists, from medical consultation in hospitals and clinics in Portugal. With the referral, it is expected that the medical doctor explains the goal and benefits of PR. Eligible patients will be contacted by the reabilitAR team, for additional questions and to begin the integration process.

Sociodemographic, anthropometric, and comorbidities; vital signs and peripheral oxygen saturation; symptoms (dyspnea, fatigue); lung function; functional capacity; exercise capacity; the impact of the disease, balance, and cognitive function will be collected before the reabilitAR program. Additionally, health care utilization will be registered.

The program consists in home visits for the exercise training and the self-management sessions, and motivational phone-calls including the follow-up of the clinical condition, the progression of exercise training, including a total of 14 home visits, with more visits in the first two weeks of the program (4 visits). From the third week, one visit will be replaced by a phone call, for a total of 10 phone calls.

After 12 weeks all outcome measures will be reassessed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD based on the GOLD criteria - postbronchodilator forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) ratio <70%;
* Electrocardiogram (ECG) record at rest;
* Written informed consent form;

Exclusion Criteria:

* Presence of any clinical condition that does not allow the participants to a home-based PR program, such as, significant cardiovascular (e.g. symptomatic ischaemic cardiac disease), neurological (e.g. neuromuscular dystrophy disease), or presence of musculoskeletal disease;
* Signs of cognitive impairment (e.g. dementia).

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-01-17 (Estimated)

PRIMARY OUTCOMES:
Change from baseline number of steps (incremental step test) at 12 weeks | At baseline and up to 12 weeks
  The incremental step test will be used to assess exercise capacity

SECONDARY OUTCOMES:
Change from baseline number of repetitions (1-minute sit-to-stand test) at 12 weeks | At baseline and up to 12 weeks
  The 1-minute sit-to-stand test will be used to assess functional capacity
Change from baseline score of CAT at 12 weeks | At baseline and up to 12 weeks
  COPD Assessment Test (CAT) will be used to assess impact of the disease. The individual score of each item is added to provide a total score that can range from 0 to 40. Total scores inferior to 10 are considered as "reduced impact", from 10-20 as "medium impact", from 21- 30 as "high impact" and above 30 as "very high impact".
Change from baseline score of dyspnea at 12 weeks | At baseline and up to 12 weeks
  Modified Borg scale will be used to assess patients' level of dyspnea. 0-10 scale is used to measure perceived dyspnea where 0 is "not at all" and 10 is "maximal"
Change from baseline score of fatigue at 12 weeks | At baseline and up to 12 weeks
  Modified Borg Scale will be used to assess patients' level of fatigue. 0-10 scale is used to measure perceived fatigue where 0 is "not at all" and 10 is "maximal"
Change from baseline score of London Chest Activities of Daily Living at 12 weeks | At baseline and up to 12 weeks
  London Chest Activities of Daily Living will be used to assess patients' level of dyspnea performing activities of daily living. The individual score of each item is added to provide a total score that can range from 0 to 75 where maximal score represents a higher level of dyspnea.
Change from baseline score of Hospital Anxiety and Depression Scale at 12 weeks | At baseline and up to 12 weeks
  Hospital Anxiety and Depression Scale will be used to assess patients' emotional status. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression symptoms.
Number of exacerbations | Up to 12 weeks
  Patients' number of hospitalizations in the previous year and during the rehabilitation will be assessed by asking the patient to self-report it.
Change from baseline score of mMRC at 12 weeks | At baseline and up to 12 weeks
  Modified British Medical Research Council (mMRC) questionnaire will be used to assess patients' level of dyspnea.This questionnaire comprises five grades in a scale from 0 to 4, with higher grades indicating greater perceived respiratory limitation.

OTHER OUTCOMES:
Short Form Berg Balance Scale 3 Point | At baseline
  Short Form Berg Balance Scale 3 Point will be used to assess patients' balance. The individual score of each item is added to provide a total score that can range from 0 to 28. Minimum score represents poor balance and maximal score represents good balance.
Mini-Mental State Examination (MMSE) | At baseline
  Mini-Mental State Examination is a 30-point questionnaire and will be used to assess patients' cognitive function. The individual score of each item is added to provide a total score that can range from 0 to 30. Total scores inferior to 9 are considered as "severe cognitive impairment", from 10-18 as "moderate cognitive impairment", from 19-23 as "mild cognitive impairment" and above 24 as "normal cognition".

CONTACTS AND LOCATIONS:
Overall Officials: Rui A Vilarinho, Master, Principal Investigator — School of Health, Polytechnic Institute of Porto
Locations (1):
- Rui Vilarinho, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Rochester CL, Vogiatzis I, Holland AE, Lareau SC, Marciniuk DD, Puhan MA, Spruit MA, Masefield S, Casaburi R, Clini EM, Crouch R, Garcia-Aymerich J, Garvey C, Goldstein RS, Hill K, Morgan M, Nici L, Pitta F, Ries AL, Singh SJ, Troosters T, Wijkstra PJ, Yawn BP, ZuWallack RL; ATS/ERS Task Force on Policy in Pulmonary Rehabilitation. An Official American Thoracic Society/European Respiratory Society Policy Statement: Enhancing Implementation, Use, and Delivery of Pulmonary Rehabilitation. Am J Respir Crit Care Med. 2015 Dec 1;192(11):1373-86. doi: 10.1164/rccm.201510-1966ST. PMID 26623686
- [Background] Bui KL, Nyberg A, Maltais F, Saey D. Functional Tests in Chronic Obstructive Pulmonary Disease, Part 1: Clinical Relevance and Links to the International Classification of Functioning, Disability, and Health. Ann Am Thorac Soc. 2017 May;14(5):778-784. doi: 10.1513/AnnalsATS.201609-733AS. PMID 28244799
- [Background] Bui KL, Nyberg A, Maltais F, Saey D. Functional Tests in Chronic Obstructive Pulmonary Disease, Part 2: Measurement Properties. Ann Am Thorac Soc. 2017 May;14(5):785-794. doi: 10.1513/AnnalsATS.201609-734AS. PMID 28244801
- [Background] Revicki D, Hays RD, Cella D, Sloan J. Recommended methods for determining responsiveness and minimally important differences for patient-reported outcomes. J Clin Epidemiol. 2008 Feb;61(2):102-9. doi: 10.1016/j.jclinepi.2007.03.012. Epub 2007 Aug 3. PMID 18177782
- [Background] Singh D, Agusti A, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Criner GJ, Frith P, Halpin DMG, Han M, Lopez Varela MV, Martinez F, Montes de Oca M, Papi A, Pavord ID, Roche N, Sin DD, Stockley R, Vestbo J, Wedzicha JA, Vogelmeier C. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease: the GOLD science committee report 2019. Eur Respir J. 2019 May 18;53(5):1900164. doi: 10.1183/13993003.00164-2019. Print 2019 May. PMID 30846476